CLINICAL TRIAL: NCT05993455
Title: A Phase 2 Basket Trial in Which Patients With Advanced Solid Tumors Carrying the KRAS G12C mUtation Receive Treatment With a Combination of Sotorasib and Panitumumab (KRAUS)
Brief Title: A Phase 2 Basket Trial in Which Patients With Advanced Solid Tumors Carrying the KRAS G12C mUtation Receive Treatment With a Combination of Sotorasib and Panitumumab
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Lee, Soo Hyeon, Associate professor, Korea University Anam Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KRAUS
Record Dates: First submitted 2023-08-03; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Efficacy
MeSH Terms: interventions — sotorasib; Panitumumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oral sotorasib + IV Panitumumab (Experimental): Oral sotorasib at a dose of 960 mg once daily with Panitumumab is administered intravenously (IV) at a dose of 6 mg/kg every 14 days, infused over 60 minutes (≤ 1,000 mg) or 90 minutes (> 1,000 mg).
  Interventions: Drug: Oral sotorasib + IV Panitumumab

INTERVENTIONS:
Drug: Oral sotorasib + IV Panitumumab — Oral sotorasib at a dose of 960 mg once daily with Panitumumab is administered intravenously (IV) at a dose of 6 mg/kg every 14 days, infused over 60 minutes (≤ 1,000 mg) or 90 minutes (> 1,000 mg).

SUMMARY:
Kirsten rat sarcoma (KRAS) mutation is one of the most common genetic mutations associated with tumor development in various human cancers, including pancreatic cancer, non-small cell lung cancer, and colorectal cancer. Previous studies have shown that KRAS mutations are present in approximately 70% of pancreatic cancer patients, 35% of colorectal cancer patients, 20% of non-small cell lung cancer patients, and 15% of cervical cancer patients. Patients with KRAS mutations generally have a shorter overall survival and increased resistance to treatment compared to wild-type tumors. KRAS mutations have been known for decades, but they have been considered "undruggable" as effective therapies targeting them were lacking.

Preclinical studies focusing on colorectal and non-small cell lung cancer cell lines have suggested that colorectal cancer cell lines exhibit a stronger response to EGFR signaling and activation of multiple RTKs (Receptor Tyrosine Kinases) than non-small cell lung cancer cell lines. As a result, they show poorer responses to KRAS G12C inhibitors, leading to the development of initial and acquired resistance to KRAS G12C inhibition. Based on this hypothesis, a phase 1-2 clinical trial, known as the KRYSTAL-1 study, was conducted in patients with metastatic colorectal cancer. The study demonstrated that the objective response rate was 19% with adagrasib monotherapy and 46% with the combination of adagrasib and cetuximab (an EGFR inhibitor), indicating that the addition of an EGFR inhibitor can overcome resistance. Building on this hypothesis, a phase 3 trial is currently underway for KRAS G12C inhibition plus EGFR blockade in metastatic colorectal cancer (ClinicalTrials.gov identifiers: NCT04793958, NCT05198934).

In this study, the aim is to investigate the efficacy of sotorasib (KRAS G12C inhibitor) plus panitumumab (EGFR inhibitor) in patients with advanced solid tumors harboring KRAS G12C mutations, who have failed standard treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have consented to participate in the KOSMOS-II observational master study.
* Age of 19 years or older.
* Histologically confirmed locally advanced or metastatic solid tumors (excluding non-small cell lung cancer and colorectal cancer) with KRAS G12C mutation detected through local next-generation sequencing analysis.
* Local advanced or metastatic disease with disease progression or unavailability of standard treatment options for the first-line anti-cancer therapy.
* Measurable lesions according to RECIST v1.1 (lesions that have not experienced disease progression after radiation therapy are excluded).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Adequate bone marrow and organ function as described below:

  ① Bone Marrow: - Absolute neutrophil count (ANC) ≥ 1,500/mm3 - Platelet count (PLT) ≥ 100,000/mm3 - Hemoglobin (Hb) ≥ 9 g/dL

  ② Liver Function:
* Total bilirubin ≤ 1.5 X upper limit of normal (ULN). If liver metastasis is present, total bilirubin up to ≤ 3 X ULN is allowed. For patients with Gilbert's syndrome, total bilirubin up to ≤ 3 X ULN and direct bilirubin within the normal range is allowed.
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 X ULN (or ≤ 5 X ULN if liver metastasis is present).

  ③ Renal Function: - Creatinine clearance ≥ 30 mL/min/1.73m2 (using the Cockcroft-Gault formula).
* Estimated life expectancy of at least 3 months according to the investigator's judgment.
* Ability to take oral medications.
* Understanding and compliance with the clinical trial protocol and ability to provide informed consent by signing the informed consent form.

Exclusion Criteria:

* Patients who have not received previous sotorasib treatment or monoclonal antibodies against epidermal growth factor receptor (EGFR) such as cetuximab or panitumumab.
* Absence of active brain metastasis or leptomeningeal metastasis (Patients with previously treated brain metastasis or leptomeningeal metastasis with radiation therapy and/or surgery [including radiosurgery] and are neurologically stable can be eligible for enrollment).
* No significant cardiovascular events within the past 6 months, such as:

.NYHA Class 3 or higher congestive heart failure. .Unstable angina or myocardial infarction. .Uncontrolled or symptomatic atrial fibrillation. .QTc prolongation (> 480 milliseconds).

* No history of stroke within the past 6 months (including transient ischemic attack).
* No diagnosis of another malignancy within 2 years prior to enrollment (excluding superficial basal cell carcinoma or squamous cell carcinoma, cervical intraepithelial neoplasia, prostate cancer under active surveillance, and well-differentiated thyroid cancer that has undergone definitive surgery).
* Pregnant or breastfeeding women.
* Participants who do not agree to effective contraception* during the clinical trial.
* Sexually active female participants of childbearing potential and their partners must agree to use medically acceptable contraception (e.g., male condoms, female condoms, or the combined use of barrier methods and spermicidal gel) during the clinical trial period and for up to 6 months after the last administration of the investigational drug.
* Male participants who have not undergone vasectomy must agree to use barrier contraception (condoms) and are prohibited from providing sperm donations until 6 months after the last administration of the investigational drug.
* Participants with active hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) infection, except under the following conditions:
* Participants who are positive for HBsAg (Hepatitis B surface antigen) can be enrolled if ALT is within the normal range and HBV DNA is <2,000 IU/ml while receiving antiviral prophylaxis for hepatitis B reactivation.
* Participants who are negative for HBsAg but positive for Hepatitis B core antibody (IgG anti-HBc) can be enrolled if HBV DNA is quantifiable but below the limit of quantification.
* Participants who are positive for anti-HCV Ab can be enrolled if HCV RNA is quantifiable but below the limit of quantification.
* Participants with planned major surgery during the clinical trial.
* Other clinically significant disorders deemed unsuitable for the clinical trial by the investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2023-09-04 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate based on RECIST v1.1 | Imaging tumor assessment time point after Cycle 1 Day 1 (each cycle is 14 days).
  Imaging tumor assessment time point after Cycle 1 Day 1 (each cycle is 14 days).

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea